CLINICAL TRIAL: NCT06751979
Title: Effect of the Probiotic Strain Streptococcus Salivarius M18 on de Novo Formation and Composition of Dental Biofilm in Orthodontic Patients: A Randomized Double-blind Placebo-controlled Clinical Trial.
Brief Title: Probiotic Treatment of Orthodontic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Bluestone Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1-10-72-77-24
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Dental Plaque; Dental Caries
MeSH Terms: conditions — Dental Plaque; Dental Caries

STUDY DESIGN:
Intervention Model Description: This clinical trial applies a randomized double-blind placebo-controlled design with two parallel arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator)
  Interventions: Dietary Supplement: Probiotic treatment
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic treatment — Daily intake of a lozenge containing the probiotic strain S. salivarius M18.
  Arms: Probiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of treatment with a lozenge containing the probiotic strain S. salivarius M18 on the formation, composition and virulence of dental plaque and in healthy orthodontic patients, compared to placebo control.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy males and females ≥ 10 years of age.
2. Able to read and receive a copy of the signed informed consent form.
3. Have at least 20 natural teeth.
4. Have been undergoing orthodontic treatment with fixed orthodontic appliances in the upper and/or lower jaw > 6 months.
5. An average plaque score of > 2 according to the Modified Orthodontic Plaque Index (MOPI) at the screening appointment.

Exclusion Criteria:

1. Significant oral soft tissue pathology based on a visual examination.
2. History of allergy or significant adverse events following use of oral hygiene products such as toothpastes, mouth rinses, breath mints, lozenges, or chewing gum or their ingredients.
3. History of allergies to milk proteins.
4. History of allergies towards probiotics.
5. Self-reported as pregnant or nursing.
6. Self-reported serious medical conditions.
7. Antibiotic or anti-inflammatory medication within 30 days of screening visit.
8. Acute sinusitis or severe oral-pharyngeal infections.
9. Smoker.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Planimetric plaque quantification | 6 weeks
  Amount of dental plaque formed after 6 weeks of probiotic treatment

SECONDARY OUTCOMES:
Prevalence of S. salivarius | Immediately after intervention
  The prevalence and abundance of S. salivarius M18 in saliva, tongue coating and dental plaque samples, as determined by 16S rRNA gene sequencing
Gingivitis | Immediately after intervention
  Gingivitis, as determined by the modified gingival index (MGI) and the sulcus bleeding index (SBI)
Plaque pH | Immediately after intervention
  The acidogenic potential of dental plaque, as determined by pH ratiometry

OTHER OUTCOMES:
Microbiome composition | Immediately after intervention
  The effects of probiotic treatment on the overall composition of the oral microbiome, assessed by next generation sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Department of Dentistry and Oral Health, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No